CLINICAL TRIAL: NCT04113746
Title: Obesity and Asthma: Unveiling Metabolic and Behavioral Pathways
Brief Title: Asthma and Obesity: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of Colorado, Denver (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Juan P Wisnivesky, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GCO 14-1859 I; R01HL129198 (NIH)
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Asthma; Obesity
Keywords: Asthma; Obesity; Self-management behaviors
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Research Coordinator who is administering the follow-up survey will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma and Exercise Lifestyle Change (Experimental): Participants receive asthma and lifestyle change education related to exercise
  Interventions: Behavioral: Better asthma self-management and incorporation of physical activity
- Asthma Education (Placebo Comparator): No lifestyle change education
  Interventions: Behavioral: Asthma Education

INTERVENTIONS:
Behavioral: Better asthma self-management and incorporation of physical activity — Participants in the asthma and exercise lifestyle change arm will participate in 4 sessions focused on behavioral change and goal-setting education to teach them how to better incorporate exercise into their daily lives and better manage their asthma. Following sessions 1 and 4, these participants will use the accelerometer to track activity, but will be blinded to the data.
  Arms: Asthma and Exercise Lifestyle Change
Behavioral: Asthma Education — General asthma education, but no discussion of the role of exercise and other lifestyle habits in asthma self-management. Following sessions 1 and 4, these participants will use the accelerometer to track activity, but will be blinded to the data.
  Arms: Asthma Education

SUMMARY:
Develop and pilot test four theory-based educational modules that integrate counseling for asthma and obesity to promote greater physical activity among people with asthma.

DETAILED DESCRIPTION:
Of the 400 obese and non-obese adult asthmatics in New York City and Denver during the 18-month observational phase of this study, the study team will randomize 80 participants (40 in NYC and 40 in Denver) into a 4-week group session pilot study focused on beliefs and behaviors associated with asthma and obesity self-management behaviors (SMB). Eligibility will be determined based on Asthma Control Questionnaire (ACQ) score and body mass index (BMI) at their 12-month visit. Participants will be randomized into an intervention or an active control arm after completing their 18-month visit. Participants will be consented into the pilot study during or after their 18-month visit. Participants will be put into groups of 7-10 for the pilot. Once formed, groups will have four 1-hour weekly visits. A person will be allowed to make up one missed session. The make-up session will be conducted on the phone or in-person depending on scheduling availability of both participant and care coach. Participants will be given accelerometers at sessions 1 and 4 that they will be asked to wear for seven days and return along with an activity diary. A follow-up survey will be administered about 30 days after the last pilot session in order to reassess the patient's asthma, obesity, exercise and medication beliefs and their adherence to asthma SMB. At the time of the follow-up survey, participants will also be given accelerometers that they will be asked to wear for seven days and return along with an activity diary.

ELIGIBILITY:
Inclusion Criteria:

* 21-64 years of age
* BMI ≥ 30
* Asthma diagnosis made by a health care provider
* Poor Asthma Control (ACQ score ≥ 0.75)
* English speaking

Exclusion Criteria:

* BMI < 30
* Good asthma control (ACQ score <0.75)
* Diagnosis of dementia
* Diagnosis of chronic obstructive pulmonary disease (COPD) or other chronic respiratory illness
* Smoking history of ≥15 pack-years owing to possible undiagnosed COPD

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P. Wisnivesky, MD, DrPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Alex D. Federman, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Fernando Holguin, MD, MPH, Principal Investigator — University of Colorado Denver, Anschutz Medical Campus
Locations (2):
- United States (2):
  - University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in May 2019 with enrollment from Oct 2019-April 2021 at Icahn School of Medicine at Mount Sinai and University of Colorado, Denver)
Groups:
- Asthma and Exercise Lifestyle Change: Participants receive asthma and lifestyle change education related to exercise
  Participants in the asthma and exercise lifestyle change arm participated in 4 sessions focused on behavioral change and goal-setting education to teach them how to better incorporate exercise into their daily lives and better manage their asthma. Following sessions 1 and 4, these participants used the accelerometer to track activity, but was blinded to the data.
- Asthma Education: No lifestyle change education
  Asthma Education: General asthma education, but no discussion of the role of exercise and other lifestyle habits in asthma self-management. Following sessions 1 and 4, these participants used the accelerometer to track activity, but was blinded to the data.
Period: Overall Study
Arm/Group | Asthma and Exercise Lifestyle Change | Asthma Education
Started | 13 | 14
Completed | 9 | 10
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asthma and Exercise Lifestyle Change | Asthma Education | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (10.7) | 48.7 (14.8) | 48 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 4 | 3 | 7
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 2 | 1 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 37 (6.5) | 39.6 (8.7) | 38.2 (7.5)
Marital Status [Count of Participants; unit: Participants]
  Married | 3 | 7 | 10
  Unmarried | 10 | 7 | 17
Language [Count of Participants; unit: Participants]
  English | 12 | 12 | 24
  Spanish | 1 | 2 | 3
Monthly Income [Count of Participants; unit: Participants]
  Less than $3000 | 9 | 10 | 19
  More than $3000 | 2 | 2 | 4
  Missing/refused | 2 | 2 | 4
Education [Count of Participants; unit: Participants]
  Elementary | 0 | 1 | 1
  Any High School | 0 | 2 | 2
  High School Graduate | 5 | 1 | 6
  Any College | 5 | 4 | 9
  College Graduate | 3 | 5 | 8
  Higher Degree | 0 | 1 | 1
Insurance [Count of Participants; unit: Participants]
  Medicare | 1 | 0 | 1
  Medicaid | 7 | 6 | 13
  Medicare and Medicaid | 0 | 1 | 1
  Private | 2 | 3 | 5
  Missing | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Beliefs About Illness Perception Questionnaire (BIPQ)
Description: BIPQ includes 5 cognitive domains (Identity, Cause, Timeline, Consequences, and Cure-Control) designed to rapidly assess the cognitive and emotional representations of illness. Each item in each domain is scored on a 0 (none) to 10 (extreme). Full scale from 0-80, where higher score reflects a more threatening view of the illness.
Time Frame: At 30 days Post-pilot follow-up visit, up to 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asthma and Exercise Lifestyle Change | Asthma Education
Number analyzed (Participants) | 9 | 10
score on a scale | 42.6 (11.4) | 36.2 (8.2)

2. Secondary Outcome: Medication Adherence Rating Scale (MARS)
Description: MARS is a self-reported questionnaire with the total score range from 0-10 with a higher score indicating better adherence.
Time Frame: At 30 days Post-pilot follow-up visit, up to 2 months
Population: Data only obtained from participants on a controller medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asthma and Exercise Lifestyle Change | Asthma Education
Number analyzed (Participants) | 7 | 9
score on a scale | 4.7 (0.5) | 4.7 (0.5)

3. Secondary Outcome: Physical Activity - Step Counts Per Day
Description: Physical activity monitoring using accelerometer and accompanying activity diary for self-report of wear. The accelerometer will measure step counts using previously determined cut-points. Based on accepted methodology, 3 or more out of the 7 days with 10 or more hours of wear time will be considered a valid measure of usual activity.
Time Frame: Week 2, Week 4, and at 30 days Post-pilot follow-up visit
Population: Data for participants with accelerometers with valid analyzable data.
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Asthma and Exercise Lifestyle Change | Asthma Education
Number analyzed (Participants) | 3 | 4
steps/day
  Week 2: number analyzed (Participants) | 1 | 4
  Week 2 | 12253.3 (0) | 2499.7 (1514.9)
  Week 4: number analyzed (Participants) | 1 | 3
  Week 4 | 13730.2 (0) | 2123.9 (1751.0)
  at 30 days post pilot follow-up visit | 2667.9 (375.4) | 3715.1 (3041.5)

4. Secondary Outcome: Time in Physical Activity
Description: Physical activity monitoring using accelerometer and accompanying activity diary for self-report of wear. The accelerometer measured time spent in different intensities of activity using previously determined cut-points. Based on accepted methodology, 3 or more out of the 7 days with 10 or more hours of wear time was considered a valid measure of usual activity.
Time Frame: Week 2, Week 4, and at 30 days Post-pilot follow-up visit
Population: Data for participants with accelerometers with valid analyzable data.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Asthma and Exercise Lifestyle Change | Asthma Education
Number analyzed (Participants) | 5 | 6
minutes/day
  Week 2: number analyzed (Participants) | 1 | 3
  Week 2 | 74.5 (0) | 8.6 (7.0)
  Week 4: number analyzed (Participants) | 1 | 3
  Week 4 | 91.5 (0) | 10.3 (8.3)
  at 30 days post pilot follow-up visit | 9.9 (6.8) | 7.8 (9.2)

5. Secondary Outcome: Asthma Control Questionnaire (ACQ)
Description: Asthma Control Questionnaire (ACQ) - self-reported asthma control validated survey, with a total score range from 0-6, with a higher score indicating severely uncontrolled asthma, used to assess current asthma control at 30 days post-pilot follow up visit.
Time Frame: at 30 days Post-pilot follow-up visit, up to 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asthma and Exercise Lifestyle Change | Asthma Education
Number analyzed (Participants) | 9 | 10
score on a scale | 1.6 (1.0) | 1.3 (0.9)

6. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ)
Description: Asthma Quality of Life Questionnaire (AQLQ) - self-reported asthma-related quality of life validated survey used to assess asthma-related quality of life at 30 days post-pilot follow-up visit. Total Score from 1-7, with higher score indicating better quality of life.
Time Frame: at 30 days post-pilot follow-up visit, up to 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asthma and Exercise Lifestyle Change | Asthma Education
Number analyzed (Participants) | 9 | 10
score on a scale | 4.9 (0.8) | 5.0 (0.6)

7. Secondary Outcome: Beliefs About Medications Questionnaire (BMQ) - Necessity and Concerns Subscale
Description: Beliefs about Medications Questionnaire (BMQ) - Necessity and Concerns
  The BMQ comprises two separate two five-item sub-scales (Necessity and Concerns) and assesses respondents' beliefs about prescribed medicines that they are currently using for specific conditions, for e.g. asthma.
  It assesses patients' beliefs about the necessity of prescribed medication for controlling their disease and their concerns about potential adverse consequences of taking it. Respondents indicate their degree of agreement with each statement on a five-point Likert scale, ranging from 1 - strongly disagree to 5 - strongly agree. Each subscale is scored from 5 -25. Scores obtained for individual items within both scales are summed. Thus, total scores for the Necessity and Concerns Scales range from 10-50. Higher scores indicate stronger beliefs in necessity or more concerns.
Time Frame: at 30 days post pilot follow-up visit, up to 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Asthma and Exercise Lifestyle Change | Asthma Education
Number analyzed (Participants) | 9 | 10
score on a scale
  Necessity Subscale | 15 (3.6) | 16.4 (5)
  Concerns Subscale | 8.4 (1) | 8.4 (2.7)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Asthma and Exercise Lifestyle Change | Asthma Education
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT04113746/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT04113746/SAP_001.pdf